CLINICAL TRIAL: NCT07162272
Title: The Efficacy of Melatonin Patches on Dental Anxiety in Children A Randomized Clinical Trial
Brief Title: The Efficacy of Melatonin Patches on Dental Anxiety in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nour Wahba, Lecturer of Pediatric Dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1512
Record Dates: First submitted 2025-07-29; First posted 2025-09-09 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Dental Anxiety; Children
Keywords: Dental Anxiety; Children; Melatonin; Melatonin Patches

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group1: Melatonin Patch (Experimental): Group 1 (n=26): Participants in the intervention group will receive two melatonin patches (each containing 1mg of melatonin, AVEELA, USA) attached to the skin of their forearm 30 minutes prior to their dental appointment according to the manufacturer's instructions. Pulse rate, blood pressure, and modified child dental anxiety scale will be measured prior to patch placement, 30minutes after their placement, after local anesthesia injection, and after completion of invasive dental treatment.
  Interventions: Drug: Melatonin Patches
- Group 2: Placebo Group (Placebo Comparator): Group 2 (n=26): The control group will receive two placebo stickers attached to the skin of their forearm at the same time point (30 minutes prior to the appointment). Pulse rate, blood pressure, and modified child dental anxiety scale will be measured prior to patch placement, 30minutes after their placement, after local anesthesia injection, and after completion of invasive dental treatment.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Drug: Melatonin Patches — Group 1 (n=26): Participants in the intervention group will receive two melatonin patches on their forearm (each containing 1mg of melatonin, AVEELA, USA) attached to the skin of their forearm 30 minutes prior to their invasive dental treatment. Pulse Rate, Blood Pressure, and Modified Child Dental Anxiety Scale will be measured before melatonin patches application, after 30minutes of patches application, then after local anesthesia injection, and finally after completing the invasive dental treatment.
  Other Names: Melatonin Stickers
  Arms: Group1: Melatonin Patch
Other: Placebo Group — Group 2 (n=26): Participants in the intervention group will receive two placebo patches on their forearm attached to the skin of their forearm 30 minutes prior to their invasive dental treatment. Pulse Rate, Blood Pressure, and Modified Child Dental Anxiety Scale will be measured before placebo patches application, after 30minutes of patches application, then after local anesthesia injection, and finally after completing the invasive dental treatment.
  Other Names: Non-melatonin patches; melatonin-free patches
  Arms: Group 2: Placebo Group

SUMMARY:
Statement of Problem:

Dental anxiety significantly impacts dental treatment outcomes, particularly in pediatric patients. Given the side effects associated with current oral anxiolytic medications, there is a need to clinically evaluate safe and natural alternatives, such as melatonin patches, to validate their efficacy.

Aim of Study:

The aim of this study is to evaluate the effect of melatonin patches on reducing dental anxiety in children. Anxiety assessments will be done by recording the pulse rate, blood pressure, and by utilization of the modified child dental anxiety scale in pediatric dental patients.

Materials and Methods:

Fifty two children will be divided into two groups. One group (n=26) will be given two melatonin patches per patient and the other group (n=26) will receive two placebo stickers 30 minutes before dental treatment. Pulse rate, blood pressure and modified child dental anxiety scale will be recorded before and after dental treatment completion as well as after the intervention for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 5-7 years old.
* Patients exhibiting Frankl's behavior rating grade III or IV.
* Children requiring invasive dental treatment in their primary teeth.

Exclusion Criteria:

* Patients with severe dental symptoms (e.g. spontaneous pain, pain not relieved by analgesics).
* History of allergy to melatonin
* Children who currently use any medication
* Orphans and special health care needs patient.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Modified Child Dental Anxiety Scale | 1 day: from recruitment to end of treatment 1 day.
  The child's anxiety will be measured using the five faces version of the modified child dental anxiety scale (MCDAS). It contains five-point Likert scale each corresponding to a smiley face that describe one of the feelings ranging from "relaxed/not worried" (1) to "very worried" (5). This will be recorded at baseline (pre-intervention), 30 minutes after melatonin patch placement (peri-operatively phase I), then immediately after local anesthesia injection (peri-operatively phase II), and immediately post-operatively.
Blood Pressure | 1 day: from recruitment to end of treatment 1 day.
  Measuring patients' systolic and diastolic blood pressure using a digital blood pressure scale. This will be recorded at baseline (pre-intervention), 30 minutes after melatonin patch placement (peri-operatively phase I), then immediately after local anesthesia injection (peri-operatively phase II), and immediately post-operatively.
Pulse rate | 1 day: from recruitment to end of treatment 1 day.
  Measuring patients' pulse rate using digital pulse oximeter scale. This will be recorded at baseline (pre-intervention), 30 minutes after melatonin patch placement (peri-operatively phase I), then immediately after local anesthesia injection (peri-operatively phase II), and immediately post-operatively.
Oxygen Saturation | 1 day: from recruitment to end of treatment 1 day.
  Measuring patients' oxygen saturation using digital pulse oximeter scale. This will be recorded at baseline (pre-intervention), 30 minutes after melatonin patch placement (peri-operatively phase I), then immediately after local anesthesia injection (peri-operatively phase II), and immediately post-operatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic of pediatric dentistry department faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided